CLINICAL TRIAL: NCT00786448
Title: Post-Marketing Surveillance Study Emselex
Brief Title: Post Marketing Surveillance Study on Emselex After Launch in Germany
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 12245; EX0501DE
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Darifenacin, Emselex (BAY79-4998)

INTERVENTIONS:
Drug: Darifenacin, Emselex (BAY79-4998) — Patients from routine practice

SUMMARY:
- Data are obtained of Emselex in routine treatment of Overactive Bladder. The general objectives are to evaluate the product safety, compatibility, efficacy and patient acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with Emselex for Overactive Bladder

Exclusion Criteria:

* Exclusion criteria are the contraindications as specified in the German product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from routine practice
Sampling Method: Non-Probability Sample
Enrollment: 5821 (Actual)
Dates: Start 2005-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Adverse events, Adverse drug reactions, physician's global assessment of tolerability | After 2-3 months of treatment (long-term 6 months)

SECONDARY OUTCOMES:
Incontinence | At end of study
Urgency episodes | At end of study
Micturitions / nycturitions | At end of study
Physician's assessment of improvement/efficacy | At end of study
Physician's assessment of patient's satisfaction with therapeutic effect | At end of study
Physician's assessment of patient's ability to hold urine | At end of study
Dose and treatment duration of Emselex | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany